CLINICAL TRIAL: NCT02735343
Title: The CHECK Trial: A Comparison of Headache Treatment in the Emergency Department: Compazine Versus Ketamine. A Multi-Center, Randomized, Double-Blind, Clinical Control Trial
Brief Title: The CHECK Trial: A Comparison of Headache Treatment in the Emergency Department: Compazine Versus Ketamine
Acronym: Check
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study goals met
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWH20160057H
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Prochlorperazine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment arm (Active Comparator): compazine 10 mg Intravenously along with diphenhydramine 25 mg Intravenously
  Interventions: Drug: Compazine
- Research arm (Experimental): Ketamine 0.3 mg/kg Intravenously along with ondansetron 4 mg Intravenously
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Compazine — Compazine 10mg with diphenhydramine 25 mg IV
  Other Names: prochlorperazine
  Arms: Standard treatment arm
Drug: Ketamine — Ketamine 0.3 mg/kg along with ondansetron 4 mg IV
  Arms: Research arm

SUMMARY:
Investigators are comparing Ketamine to prochlorperazinecompazine for benign headaches in the ED. Subjects will be randomized into 1 of 2 groups. Group 1 will receive standard treatment of prochlorperazinecompazine 10 mg IV along with diphenhydramine 25 mg IV. Group 2 (research arm) will receive Ketamine 0.3 mg/kg along with ondansetron 4 mg IV. Subjects will be seen at 15, 30, 45, and 60 minutes post-intervention to obtain Heart Rate, Blood Pressure, Headache severity, Nausea severity, Vomiting severity, Anxiety severity, and Restlessness severity. At 24-48 hours post intervention we will contact subjects and assess their pain and assess their satisfaction with their migraine pain management as part of this study. Subjects' participation will last up to 48 hours post headache.

DETAILED DESCRIPTION:
Screening Visit:

* Obtain signed Informed Consent Document and HIPAA Authorization (research-driven).
* Record: Date of birth, age, phone number, gender, race, ethnicity, social security number, name of standard of care rescue medications (over-the-counter and prescription), current email address (to be used for scheduling only), height (in inches), weight (in pounds), history of traumatic brain injury, concussion, or any mild to severe head trauma, medication use. (research only)
* Review past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) or ESSENTRIS to verify the inclusion/exclusion criteria.
* Women of childbearing potential will have a serum pregnancy test (5-10 milliliters (mls), approximately 1-2 teaspoons of blood) (research-driven).

Visit 1:

* Heart rate
* Blood pressure
* Headache severity via 100-mm VAS.
* Nausea severity via 100-mm VAS.
* Vomiting severity via 100-mm VAS.
* Anxiety severity via 100-mm VAS.
* Restlessness severity via 100-mm VAS.
* Record type and amount of rescue medications (over-the-counter and prescription) use in the past 7 days. (research only)
* Subjects will be randomized by the pharmacy. We will use a random-number generator and use blocking to ensure roughly equal sample sizes. Both subjects and investigators will be blinded to the study group assignments. Subjects will be randomized by the pharmacy into one of two groups (research-driven):

  * Group 1: Standard treatment arm (prochlorperazinecompazine 10 mg IV along with diphenhydramine 25 mg IV)
  * Group 2: Research arm (Ketamine 0.3 mg/kg along with ondansetron 4 mg IV)

    15 minutes post treatment:
* Heart rate
* Blood pressure
* Headache severity via 100-mm VAS.
* Nausea severity via 100-mm VAS.
* Vomiting severity via 100-mm VAS.
* Anxiety severity via 100-mm VAS.
* Restlessness severity via 100-mm VAS.

  30 minutes post treatment:
* Heart rate
* Blood pressure
* Headache severity via 100-mm VAS.
* Nausea severity via 100-mm VAS.
* Vomiting severity via 100-mm VAS.
* Anxiety severity via 100-mm VAS.
* Restlessness severity via 100-mm VAS.

  45 minutes post treatment:
* Heart rate
* Blood pressure
* Headache severity via 100-mm VAS.
* Nausea severity via 100-mm VAS.
* Vomiting severity via 100-mm VAS.
* Anxiety severity via 100-mm VAS.
* Restlessness severity via 100-mm VAS.

  60 minutes post treatment:
* Heart rate
* Blood pressure
* Headache severity via 100-mm VAS.
* Nausea severity via 100-mm VAS.
* Vomiting severity via 100-mm VAS.
* Anxiety severity via 100-mm VAS.
* Restlessness severity via 100-mm VAS.

24-48 hours post treatment:

* Subjects will be contacted either in-person or via phone and the following information will be collected:

  * Subjects will be asked "On a scale of 0-10, with 10 being the worst pain, what is your current level of pain?"
  * Subjects will be asked "On a scale of 0 to 10, how satisfied were you with you're the migraine pain management as part of this research study? (dissatisfied 0 - 10 very satisfied)
* Subjects will be alerted to what group they were randomized into.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion Criteria

* Age 18 to 65 years who present to the ED with complaint of a headache
* Temperature less than 100.4 F
* Diastolic blood pressure less than 104 mm Hg
* Normal neurologic exam and normal mental status

Exclusion Criteria

* Pregnant or breastfeeding
* Meningeal signs are present
* Acute angle closure glaucoma is suspected
* Head trauma within the previous two weeks
* Lumbar puncture within the previous two weeks
* Thunderclap (rapid) onset of the headache
* Weight more than 150 kg or less than 40 kg
* Known allergy to diphenhydramine
* Known allergy to ondansetron. (Zofran)
* Known allergy to Compazine
* Known allergy to Ketamine
* History of schizophrenia or bipolar disorder
* History of intracranial hypertension
* Is a prisoner
* Patient declined informed consent
* Non-English speaking patient
* Attending provider excludes patient
* Elderly patients with dementia
* Patients with severe headaches that diminish their decision making capability will not be able to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pitotti, MD, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with University Medical Center of Southern Nevada via a Cooperative Research and Development Agreement. They are conducing the same study under a different IRB.

REFERENCES:
- [Derived] Driver BE, Klein LR, Carlson K, Harrington J, Reardon RF, Prekker ME. Preoxygenation With Flush Rate Oxygen: Comparing the Nonrebreather Mask With the Bag-Valve Mask. Ann Emerg Med. 2018 Mar;71(3):381-386. doi: 10.1016/j.annemergmed.2017.09.017. Epub 2017 Oct 28. PMID 29089172
- [Derived] Zitek T, Gates M, Pitotti C, Bartlett A, Patel J, Rahbar A, Forred W, Sontgerath JS, Clark JM. A Comparison of Headache Treatment in the Emergency Department: Prochlorperazine Versus Ketamine. Ann Emerg Med. 2018 Mar;71(3):369-377.e1. doi: 10.1016/j.annemergmed.2017.08.063. Epub 2017 Oct 14. PMID 29033296

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Treatment Arm | Research Arm
Started (study was terminated as no longer necessary) | 1 | 4
Completed | 1 | 2
Not Completed | 0 | 2
Not completed — screen fail | 0 | 2

BASELINE CHARACTERISTICS:
Population: This study was terminated early due to the study becoming unnecessary due to findings in another trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Arm | Research Arm | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 3 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Subjects marked a line on a Visual Analogue Scale rating from None to Severe. Study staff measured the mark in millimeters and converted to a scale from 0 to 100 possible points, with 100 being most severe.
Time Frame: 15 min, 30 min, 45 min, 60 min
Population: This study was terminated early due to the study becoming unnecessary due to findings in another trial. Raw data were collected for the 3 subjects who completed the study (2 screen failed). Raw data is reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Standard Treatment Arm | Research Arm
Number analyzed (Participants) | 1 | 2
score on a scale
  Headache Score 0 minutes | 39 [39 to 39] | 74 [68 to 80]
  headache score 15 minutes | 18 [18 to 18] | 16.5 [16 to 17]
  headache score 30 minutes: number analyzed (Participants) | 1 | 1
  headache score 30 minutes | 8 [8 to 8] | 19 [NA to NA] — 1 subject lost to followup. The remaining subject scored 19.
  headache score 45 minutes: number analyzed (Participants) | 0 | 1
  headache score 45 minutes |  | 10 [NA to NA] — 1 subject lost to followup. The remaining subject scored 10.
  headache score 60 minutes: number analyzed (Participants) | 0 | 1
  headache score 60 minutes |  | 13 [NA to NA] — 1 subject lost to followup. The remaining subject scored 13.

ADVERSE EVENTS:
Time Frame: This study was terminated early due to the study becoming unnecessary due to findings in another trial. 5 subjects were enrolled before termination and were followed until they had completed the study, 48 hours post treatment.
Description: This study was terminated early due to the study becoming unnecessary due to findings in another trial. 5 subjects were enrolled before termination and were followed until they had completed the study, 48 hours post treatment.
Arm/Group | Standard Treatment Arm | Research Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
This study was terminated early due to the study becoming unnecessary due to findings in another trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT02735343/Prot_SAP_000.pdf